CLINICAL TRIAL: NCT01807741
Title: Asenapine for Bipolar Depression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding ended due to recruitment delays
Sponsor: University of Cincinnati (Other)
Collaborators: University of Louisville (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Caleb M. Adler, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-4181
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Bipolar Depression
Keywords: Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — asenapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine Group (Experimental): Asenapine will be given beginning on day 0 at 5 mg bid. Dose will be increased to 10 mg bid if there is less than 50% decrease in MADRS score by week 2. Dose increases may be held if clinically indicated. Doses may be decreased at any time, if clinically indicated, by increments of 5 mg/day to a minimum of 5 mg qHS. Daily treatment with asenapine will be for 8 weeks.
  Interventions: Drug: Asenapine
- Placebo Group (Active Comparator): Sublingual tablets similar to the asenapine tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Available in 5 and 10 mg.
  Other Names: Saphris
  Arms: Asenapine Group
Drug: Placebo
  Other Names: sugar pill
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to compare asenapine with placebo in the treatment of depression associated with bipolar disorder, type I over eight weeks.

We hypothesize that patients will show significantly greater improvement with asenapine than placebo over eight weeks of treatment.

DETAILED DESCRIPTION:
86 patients with an episode of major depression associated with bipolar disorder, type I will be recruited by two sites for the study over fifteen months. Medication will be administered in a double-blind manner. Patients will receive asenapine (or placebo) beginning on day 0 at 5 mg bid. Dose may be increased to 10 mg bid and adjusted based on clinical response. Patients will be evaluated by a blinded (to treatment status) rater. Patients will be seen and ratings obtained at baseline (day 0) and on days 7, 14, 28, 42, and 56 (or termination from the study). Adverse events will be evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for bipolar depression based on the MINI and confirmation of a previous manic or mixed episode
* 18-55 years of age
* Female patients must be using a medically accepted means of contraception (e.g. oral contraceptives, Depo-Provera, abstinence)
* Each patient must understand the nature of the study and must provide written informed consent
* Patients must have a diagnosis of bipolar disorder, type I and currently display an acute depressive episode as determined by M.I.N.I. (Sheehan et al, 1998)
* Patients must have a baseline (day 0) MADRS score ≥26
* Current episode of depression must have persisted for at least one month and no more than six months at study entry
* Subjects should be fluent in English

Exclusion Criteria:

* Female patients who are either pregnant or lactating
* Clinically significant or unstable hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions
* Any history of current or past diabetes that was treated with pharmacological intervention
* Neurological disorders including epilepsy, stroke, or severe head trauma
* Clinically significant laboratory abnormalities, on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, lipid profile, fasting glucose, urinalysis, thyroid indices and EKG
* Depression due to a general medical condition or substance-induced depression (DSM-IV)
* Mental retardation (IQ <70)
* Meeting criteria for a mixed episode, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* History of hypersensitivity to or intolerance of asenapine
* Prior history of asenapine non-response
* DSM-IV substance (except nicotine or caffeine) dependence within the past 3 months
* Judged clinically to be at suicidal risk (defined as having active suicidal ideation, intent or plan, or a serious suicide attempt within 30 days, or a baseline MADRS suicide score of >4)
* Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry
* Failure of the current depressive episode to respond to two or more pharmacological interventions
* Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0
* Schizophrenia or other psychotic disorders (including schizophreniform disorder, schizoaffective disorder, delusional disorder, brief psychotic disorder, shared psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV
* Major depressive disorder, dysthymic disorder, depressive disorder not otherwise specified

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Depression Score | 8 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS)will be used as a measure of efficacy reflecting change in MADRS total scores from baseline to endpoint over 8 weeks.

SECONDARY OUTCOMES:
Change in Depression Response Rate | 8 weeks
  MADRS Response Rate: Defined by a ≥ 50% decrease from baseline to endpoint in MADRS total score over 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Caleb M Adler, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States